CLINICAL TRIAL: NCT02894151
Title: Effectiveness of Levonorgestrel-intrauterine System (LNG-IUS) Versus Depot Medroxyprogesterone Acetate (DMPA) in Treatment of Pelvic Pain in Clinically Diagnosed Endometriotic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 523/57
Record Dates: First submitted 2016-08-31; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Clinically Diagnosed Endometriotic Patient Was Defined as a Woman Who Has Pelvic Pain and at Least One Evidence of PV or TVS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LNG-IUS (Active Comparator): LNG IUS was hormonal containing IUD relased LNG at constant rate through out 5 year period.
  It was inserted only first time entry in the study.
  Interventions: Device: LNG-IUS
- DMPA (Active Comparator): DMPA was given in trimonthly intramuscular injection.
  Interventions: Drug: Depot medroxyprogesterone acetate

INTERVENTIONS:
Drug: Depot medroxyprogesterone acetate
  Arms: DMPA
Device: LNG-IUS
  Arms: LNG-IUS

SUMMARY:
The primary objective : To compare effectiveness of pain control in endometriosis associated pelvic pain between LNG-IUS and DMPA The secondary objective : To compare vaginal bleeding pattern, side effect, continuation rate, satisfaction and quality of life between LNG-IUS and DMPA in treatment of endometriosis associated pelvic pain

DETAILED DESCRIPTION:
The participants were randomized into two treatment groups, by Block Of Four method, LNG-IUS and DMPA group. For the patients in the LNG-IUS group, a LNG-IUS (Mirena) was inserted. The system released the active ingredient LNG for up to five years at a virtually constant rate. For the patients in the Depot MPA Group, 150 mg depot MPA was given intramuscularly once every three months.

All participants were recieved the individual calendars to record all vaginal bleeding occured during treatment. The amount of bleeding was described relative to normal menstruation of each patient; less than, same as, more than their baseline menses. To use easily, we assigned the symbols to represent quantity of vaginal bleeding as described. Each symbol was recorded every day except no bleeding, which was represented with blank space in the calendar. The bleeding pattern were assessed as bleeding rating score; less than normal menses = 1, same amount of normal menses = 2, more than normal menses = 3. No bleeding was defined as 30 consecutive days with bleeding score 0. The mean bleeding score was calculated by sum of the daily scores in each month period.

Follow-up visits were scheduled three times at months 1, 3 and 6 after initial treatment. At each visit, VAS and bleeding pattern was recorded. Side-effects of the two therapies were checked. Patients were allowed to choose to withdraw from their designated therapy at any time. The follow-up was completed in May 2016 for the last patient.

At the final visit, 6 months after treatment, all participants in both treatment groups were recorded the datas of blood pressure, body weight, transvaginal ultrasonography, lipid profiles and SF-36 quesionaires. In addition, all50 patients were asked whether they want to continue in the given treatement and the reason of discontinuation including the satisfaction scores during therapy were rated as 1-5 Likert-scale; 1-very dissatisfied, 2- dissatisfied, 3-neither satisfied/dissatisfied, 4-satisfied, 5-very satified.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45year Pelvic pain VAS>50 Previous Sexual intercouse

Exclusion Criteria:

* other genital tract disease causing pelvic pain Previous hromonal treament 3 month History of DMPA treatment failure WHO eligibility criteria 2009 categorized in 3-4 for DMPA and LNG-IUS user Fertility desire within 1 year Psychoneurosis Pregnant and breast fed women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change baseline pain score assessed by visual analog scale after 6 month-use of both interventions | 1year